CLINICAL TRIAL: NCT05114772
Title: Pre Procedural High Serum Visfatin and Tumor Necrosis Factors "Alpha" Might Predict Recurrent Atrial Fibrillation After Catheter Ablation
Brief Title: Pre Procedural Biomarkers Might Predict Recurrent Atrial Fibrillation After Catheter Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Fayez Al-kassas, lecturer of Cardiology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 34816/7/19
Record Dates: First submitted 2021-10-01; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recurrent Atrial fibrillation (Active Comparator): patients developed Recurrent Atrial fibrillation catheter ablation
  Interventions: Diagnostic Test: Measuring Serum bio-markers
- NO Recurrent Atrial fibrillation (Active Comparator): patients didn't develop Recurrent Atrial fibrillation catheter ablation
  Interventions: Diagnostic Test: Measuring Serum bio-markers

INTERVENTIONS:
Diagnostic Test: Measuring Serum bio-markers — ELISA Estimation of Serum visfatin and tumor necrosis factor-alpha

SUMMARY:
Evaluation of the predictive value of serum levels of adipocytokines and primary phase reactant for recurrent atrial fibrillation (RAF) after catheter ablation in 26 patients had persistent and 91 patients had paroxysmal AF. During 12-m follow-up, 41 patients had RAF (35%). Patients had RAF were significantly older, had significantly higher BMI, lower ejection fraction and wider maximal left atrial diameter (LAD). Serum hs-CRP, IL-6, TNF-α, visfatin, and adiponectin levels were significantly higher in patients developed. Elevated serum levels of TNF-α, visfatin and adiponectin are a significant positive predictors for RAF.

DETAILED DESCRIPTION:
Objectives: Estimation of serum levels of visfatin, adiponectin, tumor necrosis factor-α (TNF-α), interleukin-6 (IL-6) and high-sensitivity C-reactive protein (hs-CRP) in patients had atrial fibrillation (AF) resistant to medical treatment and assigned to catheter ablation (CA) to evaluate these biomarkers as predictors for recurrent AF (RAF).

Patients & Methods: 117 patients; 26 patients had persistent and 91 patients had paroxysmal AF underwent had clinical and echographic evaluations and gave blood samples for ELISA estimation of serum levels of studied cytokines. CA was performed through isolation of all pulmonary veins according to the stepwise procedure of ablation. Patients were re-evaluated every three months till 12-m follow-up for post-procedural RAF.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal or persistent AF that was resistant to medical acceptable daily dose therapy in patients who were free of exclusion criteria and accepted to sign the written fully informed consent to undergo CA and to give pre-procedural blood samples.

Exclusion Criteria:

* History of the presence of longstanding persistent or permanent AF,
* myocardial infarction, acute coronary syndrome (ACS),
* significant heart failure (NYHA3),
* dilated or hypertrophic cardiomyopathy,
* left ventricular ejection fraction (LVEF)< 35%, congenital pathologies,
* significant valvular heart disease,
* pulmonary embolism,
* venous thrombosis,
* intracardiac thrombus or inability to take warfarin or other oral anticoagulants,
* hepatic or renal insufficiency,
* acute inflammatory states (sepsis, chronic obstructive pulmonary disease in acute phase),
* cancer,
* autoimmune pathologies.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Recurrent Atrial Fibrillation | 12 months
  Recurrent Atrial Fibrillation after Catheter ablation

CONTACTS AND LOCATIONS:
Overall Officials: Amr El kassas, MD, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Egypt